CLINICAL TRIAL: NCT06606938
Title: Faecal Microbiota Transplantation for Insomnia Disorder: a Randomized, Double-blind, Placebo-controlled Trial
Brief Title: FMT for Insomnia Disorder (FMT-SLEEP)
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Siew Chien NG, Professor Siew Chien NG, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FMT-SLEEP
Record Dates: First submitted 2024-08-23; First posted 2024-09-23 (Actual); Last update posted 2024-09-23 (Actual); Status verified 2024-09

CONDITIONS: Chronic Insomnia Disorder
Keywords: Faecal Microbiota Transplantation
MeSH Terms: interventions — Fecal Microbiota Transplantation; Saline Solution

STUDY DESIGN:
Intervention Model Description: The intervention group will receive FMT while the control group will receive 0.9% sodium chloride solution (normal saline) as placebo.
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Faecal Microbiota Transplantation (Experimental): FMT will be reconstituted from healthy donor's stool
  Interventions: Procedure: Faecal Microbiota Transplantation
- Placebo (Sham Comparator): Subjects will receive 0.9% sodium chloride solution (normal saline) as placebo identical looking with FMT
  Interventions: Procedure: Normal Saline (Placebo)

INTERVENTIONS:
Procedure: Faecal Microbiota Transplantation — FMT at baseline, week 2, week 4
  Arms: Faecal Microbiota Transplantation
Procedure: Normal Saline (Placebo) — Placebo at baseline, week 2, week 4
  Arms: Placebo

SUMMARY:
Insomnia disorder is characterized by difficulty initiating or maintaining sleep, or early morning awakening accompanied by symptoms such as irritability or fatigue during wakefulness. It is one of the most prevalent health concerns in the population and in clinical practice, with more than one-third of adults experience transient insomnia at some point in their lives. In about 40% of cases, insomnia can develop into a more chronic condition. The COVID-19 pandemic has further aggravated sleep problems, with a reported global prevalence of sleep disturbances reaching 40-49%. The implications of insomnia disorder are substantial, encompassing social, economic, psychological, and physical aspects.

Behavioural, cognitive, and pharmacological interventions can all be effective for insomnia. Pharmacological treatment is commonly used but may have drawbacks such as adverse events and inconclusive safety data for certain medications. Many licensed drugs can be effective in the acute treatment of insomnia but are associated with poor tolerability, or information about long-term effects is not available. Alternatively, cognitive behavioural therapy for insomnia (CBT-I), has been recommended as the first-line treatment for chronic insomnia in adults of any age according to the American and European guidelines. But issue of accessibility, compliance/adherence, and moderate response limit the practicality and applicability of CBT-I.

Recent evidence suggests that the gut microbiota plays a role in regulating sleep behaviour, both directly and indirectly. This has led to the exploration of gut microbiota modulation as a potential therapy for insomnia. Faecal microbiota transplantation (FMT), which is the infusion of faeces from healthy donors to the gut of affected subjects, has shown impressive therapeutic effects for various diseases. Several real-world studies have demonstrated improvements in symptoms of insomnia disorder following FMT. One previous study also indicated the potential of FMT in alleviating post-COVID insomnia. In this randomised, double-blind, placebo-controlled trial, the investigators aim to assess the efficacy of FMT in improving insomnia disorder. Two groups will be recruited in 1:1 ratio. The intervention group will receive FMT while the control group will receive normal saline as placebo. Both groups will have the same assessments.

DETAILED DESCRIPTION:
Insomnia disorder is characterized by difficulty initiating or maintaining sleep, or early morning awakening accompanied by daytime symptoms such as irritability or fatigue. It is one of the most prevalent health problems in the population and in clinical practice, with more than one-third of adults experience transient insomnia at some point in their lives. In about 40% of cases, insomnia can develop into a more chronic condition. The COVID-19 pandemic has further aggravated sleep problems, with a reported global prevalence of sleep disturbances reaching 40-49%. The social, economic, psychological and physical implications of insomnia disorder are substantial, with evidence linking the condition to an increased risk of hypertension, cardiovascular disease, anxiety, and depression, as well as impaired quality of life, work absenteeism, work-related accidents, poor work efficiency, and family dysfunction.

Behavioural, cognitive, and pharmacological interventions can all be effective for insomnia. Pharmacological treatment is common in practice and widely used for the management of insomnia. A recent meta-analysis suggested that Eszopiclone and Lemborexant had the best profile in terms of efficacy, acceptability, and tolerability. However, Eszopiclone might cause substantial adverse events and safety data on lemborexant were inconclusive. Many licensed drugs (including benzodiazepines, Z-hypnotics and dual orexin receptor antagonist, DORA) are prescribed as effective short-term treatment of insomnia but some are associated with poor tolerability, or the information about long-term safety effects is not available. Alternatively, cognitive behavioral therapy for insomnia (CBT-I), has been recommended as the first-line treatment for chronic insomnia in adults of any age according to the American and European guidelines. But issues of accessibility, compliance/adherence, and moderate response also pose limit the practicality and applicability of CBT-I.

Growing evidence indicates that the microbiota-gut-brain axis contributes to the regulation of sleep behavior both directly and indirectly and may play a critical role in the etiology and pathogenesis of sleep disorders. Sleep loss is capable of altering the gut microbiota composition through increased hunger and decreased physical activity, immunomodulation, or hypothalamus-pituitary-adrenal (HPA) axis activation and subsequent intestinal barrier disruption. Conversely, the gut microbiome is capable of altering sleep through somnogenic lipopolysaccharide (LPS) and Muramyl peptides translocation, vagal afferent excitation in response to enteric LPS, regulation of enterochromaffin cell serotonin production, and inflammatory cytokine regulation. Consequently, gut microbiota modulation is a potential therapy for insomnia.

According to a preclinical study, transplantation of the gut microbiota from mice with sleep disorder into normal mice induced microglia overactivation and neuronal apoptosis in the hippocampus, cognitive decline, and colonic microbiota disorder. Moreover, a human study found that fecal microbiota transplantation (FMT) from healthy donors improved sleep and also ameliorated depression and anxiety in patients with irritable bowel syndrome (IBS). Another study demonstrated that FMT led to a decrease in the scores of the five components of Pittsburgh Sleep Quality Index (PSQI) in 52 IBS patients with poor sleep quality, including subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, and sleep disturbances. A clinical study showed significantly lower Sleep Disturbance Scale for Children (SDSC) scores in children with autism after FMT, whilst a retrospective study also indicated that FMT could significantly improve the sleep disorder scores in the autistic children with constipation. According to a real world study, FMT significantly ameliorated the Insomnia Severity Index (ISI), Pittsburgh Sleep Quality Index (PSQI), and quality of life in patients with chronic insomnia. The results from one previous study also demonstrated that FMT could alleviate post-COVID insomnia.

In this randomised, double-blind, placebo-controlled trial, the investigators aim to assess the efficacy of FMT in improving insomnia disorder. The investigators hypothesize that FMT is a safe and effective treatment for insomnia disorder.

ELIGIBILITY:
Inclusion Criteria:

* 1. Individuals aged 18 and above
* 2. Subjects who were diagnosed with chronic insomnia disorder according to the Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5) and with moderate or above insomnia disorder defined as ISI > 14

Exclusion Criteria:

* 1. Having an additional sleep disorder, such as restless legs syndrome, or circadian rhythm sleep disorder, that can significantly disrupt the sleep cycle as ascertained by Diagnostic Interview for Sleep Patterns and Disorders (DISP)
* 2. Requiring immediate psychiatric care (e.g., imminently suicidal subjects) or have attempted suicide in the past 6 months
* 3. Change of treatment or therapy for insomnia within 4 weeks
* 4. Known history of severe organ failure (including decompensated cirrhosis), renal failure on dialysis, suffering from human immunodeficiency virus infection
* 5. Confirmed active malignancy
* 6. Had abdominal surgery
* 7. Contraindications to GI endoscopy
* 8. On shift work
* 9. Taking antibiotics, probiotic or prebiotic preparations within 4 weeks
* 10. Known pregnancy
* 11. Mental retardation or inability to provide informed consent
* 12. Are participating in other interventional studies

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Estimated)
Dates: Start 2024-11-01 (Estimated); Primary Completion 2026-10-31 (Estimated); Study Completion 2027-04-30 (Estimated)

PRIMARY OUTCOMES:
Proportion of subjects in remission | week 8
  Proportion of subjects in remission (Insomnia Severity Index (ISI) < 8) by week 8. ISI is a self-report questionnaire used to evaluate the nature, severity and impact of insomnia. Total score ranges from 0 to 28. Higher score indicates more severe insomnia

SECONDARY OUTCOMES:
Proportion of subjects in remission | weeks 2, 4, and 24
  Proportion of subjects in remission (Insomnia Severity Index (ISI) below 8)
Proportion of subjects with response | weeks 2, 4, 8, and 24
  Proportion of subjects with response of a reduction of ISI above 6
Change in anxiety symptoms | weeks 2, 4, 8, and 24
  Anxiety symptoms will be assessed by a 7-item Generalised Anxiety Disorder-7 scale (GAD-7). GAD-7 is a widely used diagnostic self-report scale for the screening, diagnosis and severity assessment of anxiety disorder. Total score ranges from 0 to 21. Higher score indicates more severe anxiety.
Change in depression symptoms | weeks 2, 4, 8, and 24
  Depresion symptoms will be evaluated by the Patient Health Questionnaire-9 (PHQ-9), a 9-item instrument. Total score categories for PHQ-9 are: 0-4 = Minimal/no depression, 5-9 = Mild depression, 10-14 = Moderate depression, 15-19 = Moderately severe depression, 20-27 = Severe depression.
Change in daytime sleepiness | weeks 2, 4, 8, and 24
  Daytime sleepiness will be measured by using the Epworth Sleepiness Scale (ESS). The ESS consists of eight situations in which individuals rate their likelihood of nodding off on a scale of 0 to 3, where 0 represents "Would Never Nod Off" and 3 represents "High Chance of Nodding Off". To obtain a total score on the ESS, the scores for each of the eight situations are summed, resulting in a range from 0 to 24. Higher scores indicate a higher level of daytime sleepiness.
Change in sleep efficiency by actigraph | weeks 8 and 24
  Actigraph is a non-invasive method used to monitor and measure activity levels and sleep patterns over a period. It contains an accelerometer that measures activity and provides data on the intensity, duration, and frequency of physical movements. Sleep and wake status will be determined by algoraithm that calculate activity count measured by the accelerometer. Bedtime, wakeup time, sleep duration, sleep onset latency and sleep efficiency will be generated.
Change in sleep pattern by sleep diary | weeks 2, 4, 8, and 24
  The Sleep Diary is also utilised to record the quality and quantity of subjects' sleep. A sleep diary is a tool used to track and record various aspects of an individual's sleep patterns and habits over a period of time. It provides a detailed account of sleep-related information that can be helpful for assessing sleep quality, identifying patterns or issues, and guiding treatment or behavior modifications. The sleep diary will include the following information: Date, Bedtime, Sleep onset, Wake-up time, Sleep duration, Number of awakenings, Sleep quality, Napping, and Comments.
Change in Patient Global Impression - Improvement | weeks 2, 4, 8, and 24
  The Patient Global Impression-Improvement (PGI-I) will be used to assess subjects' perceptions regarding the effects of study invention on their sleep. The PGI-I scale consists of a single question that asks the patient to rate their improvement since the start of the study invention, using a seven-point scale ranging from very much improved to very much worse.
Change in quality of life | weeks 8, and 24
  The quality of life of subjects will be evaluated via 12-item Short Form Survey (SF-12) covering eight domains: Limitations in physical activities because of health problems; Limitations in social activities because of physical or emotional problems; Limitations in usual role activities because of physical health problems; Bodily pain; General mental health (psychological distress and well-being); Limitations in usual role activities because of emotional problems; Vitality (energy and fatigue); General health perceptions. The SF-12 provides two summary scores: the Physical Component Summary (PCS) score and the Mental Component Summary (MCS) score. Both summary scores are calculated based on a standardized scoring algorithm, which assigns weights to each of the 12 items and combines the responses to generate a score. A higher PCS score suggests better physical health functioning and a higher MCS score represents better mental health.
Change in fatigue scale | weeks 2, 4, 8, and 24
  The Multidimensional Fatigue Inventory (MFI) will be used to evaluate subjects' fatigue. The MFI is a 20-item scale designed to evaluate five dimensions of fatigue: general fatigue, physical fatigue, reduced motivation, reduced activity, and mental fatigue. For each item, subjects rate their experience of fatigue on a scale, ranging from 1 to 5. Higher scores indicate higher levels of fatigue within each subscale. The total score for each subscale is typically obtained by summing the scores of the corresponding items.
Change in sleep-related beliefs and attitudes | weeks 2, 4, 8, and 24
  Subjects' beliefs and attitudes towards sleep will be assessed by the Dysfunctional Beliefs and Attitudes About Sleep Scale (DBAS)-16. Subjects rate their agreement with each item on a Likert scale, ranging from 1 to 10. Higher scores indicate a greater presence of dysfunctional beliefs and attitudes related to sleep.
Change in gut microbiota composition | week 8
  Relative abundance of gut microbiota at species level will be assessed by metagenomic analysis.
Change in mucosal microbiota composition | week 4
  Relative abundance of mucosal microbiota at species level will be assessed by metagenomic analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Siew Chien Ng, PhD,FRCP, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Prince of Wales Hospital, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Buysse DJ. Insomnia. JAMA. 2013 Feb 20;309(7):706-16. doi: 10.1001/jama.2013.193. PMID 23423416
- [Background] K Pavlova M, Latreille V. Sleep Disorders. Am J Med. 2019 Mar;132(3):292-299. doi: 10.1016/j.amjmed.2018.09.021. Epub 2018 Oct 4. PMID 30292731
- [Background] Jahrami HA, Alhaj OA, Humood AM, Alenezi AF, Fekih-Romdhane F, AlRasheed MM, Saif ZQ, Bragazzi NL, Pandi-Perumal SR, BaHammam AS, Vitiello MV. Sleep disturbances during the COVID-19 pandemic: A systematic review, meta-analysis, and meta-regression. Sleep Med Rev. 2022 Apr;62:101591. doi: 10.1016/j.smrv.2022.101591. Epub 2022 Jan 22. PMID 35131664
- [Background] Sivertsen B, Lallukka T, Salo P, Pallesen S, Hysing M, Krokstad S, Simon Overland. Insomnia as a risk factor for ill health: results from the large population-based prospective HUNT Study in Norway. J Sleep Res. 2014 Apr;23(2):124-32. doi: 10.1111/jsr.12102. PMID 24635564
- [Background] Grandner MA. Sleep, Health, and Society. Sleep Med Clin. 2022 Jun;17(2):117-139. doi: 10.1016/j.jsmc.2022.03.001. Epub 2022 Apr 22. PMID 35659068
- [Background] Taddei-Allen P. Economic burden and managed care considerations for the treatment of insomnia. Am J Manag Care. 2020 Mar;26(4 Suppl):S91-S96. doi: 10.37765/ajmc.2020.43008. PMID 32282179
- [Background] Leger D, Bayon V. Societal costs of insomnia. Sleep Med Rev. 2010 Dec;14(6):379-89. doi: 10.1016/j.smrv.2010.01.003. Epub 2010 Mar 31. PMID 20359916
- [Background] Leach MJ, Page AT. Herbal medicine for insomnia: A systematic review and meta-analysis. Sleep Med Rev. 2015 Dec;24:1-12. doi: 10.1016/j.smrv.2014.12.003. Epub 2014 Dec 17. PMID 25644982
- [Background] Pan B, Ge L, Lai H, Hou L, Tian C, Wang Q, Yang K, Lu Y, Zhu H, Li M, Wang D, Li X, Zhang Y, Gao Y, Liu M, Ding G, Tian J, Yang K. The Comparative Effectiveness and Safety of Insomnia Drugs: A Systematic Review and Network Meta-Analysis of 153 Randomized Trials. Drugs. 2023 May;83(7):587-619. doi: 10.1007/s40265-023-01859-8. Epub 2023 Mar 22. PMID 36947394
- [Background] De Crescenzo F, D'Alo GL, Ostinelli EG, Ciabattini M, Di Franco V, Watanabe N, Kurtulmus A, Tomlinson A, Mitrova Z, Foti F, Del Giovane C, Quested DJ, Cowen PJ, Barbui C, Amato L, Efthimiou O, Cipriani A. Comparative effects of pharmacological interventions for the acute and long-term management of insomnia disorder in adults: a systematic review and network meta-analysis. Lancet. 2022 Jul 16;400(10347):170-184. doi: 10.1016/S0140-6736(22)00878-9. PMID 35843245
- [Background] Qaseem A, Kansagara D, Forciea MA, Cooke M, Denberg TD; Clinical Guidelines Committee of the American College of Physicians. Management of Chronic Insomnia Disorder in Adults: A Clinical Practice Guideline From the American College of Physicians. Ann Intern Med. 2016 Jul 19;165(2):125-33. doi: 10.7326/M15-2175. Epub 2016 May 3. PMID 27136449
- [Background] Riemann D, Espie CA, Altena E, Arnardottir ES, Baglioni C, Bassetti CLA, Bastien C, Berzina N, Bjorvatn B, Dikeos D, Dolenc Groselj L, Ellis JG, Garcia-Borreguero D, Geoffroy PA, Gjerstad M, Goncalves M, Hertenstein E, Hoedlmoser K, Hion T, Holzinger B, Janku K, Jansson-Frojmark M, Jarnefelt H, Jernelov S, Jennum PJ, Khachatryan S, Krone L, Kyle SD, Lancee J, Leger D, Lupusor A, Marques DR, Nissen C, Palagini L, Paunio T, Perogamvros L, Pevernagie D, Schabus M, Shochat T, Szentkiralyi A, Van Someren E, van Straten A, Wichniak A, Verbraecken J, Spiegelhalder K. The European Insomnia Guideline: An update on the diagnosis and treatment of insomnia 2023. J Sleep Res. 2023 Dec;32(6):e14035. doi: 10.1111/jsr.14035. PMID 38016484
- [Background] Riemann D, Baglioni C, Bassetti C, Bjorvatn B, Dolenc Groselj L, Ellis JG, Espie CA, Garcia-Borreguero D, Gjerstad M, Goncalves M, Hertenstein E, Jansson-Frojmark M, Jennum PJ, Leger D, Nissen C, Parrino L, Paunio T, Pevernagie D, Verbraecken J, Weess HG, Wichniak A, Zavalko I, Arnardottir ES, Deleanu OC, Strazisar B, Zoetmulder M, Spiegelhalder K. European guideline for the diagnosis and treatment of insomnia. J Sleep Res. 2017 Dec;26(6):675-700. doi: 10.1111/jsr.12594. Epub 2017 Sep 5. PMID 28875581
- [Background] Lau RI, Su Q, Ching JYL, Lui RN, Chan TT, Wong MTL, Lau LHS, Wing YK, Chan RNY, Kwok HYH, Ho AHY, Tse YK, Cheung CP, Li MKT, Siu WY, Liu C, Lu W, Wang Y, Chiu EOL, Cheong PK, Chan FKL, Ng SC. Fecal Microbiota Transplantation for Sleep Disturbance in Post-acute COVID-19 Syndrome. Clin Gastroenterol Hepatol. 2024 Dec;22(12):2487-2496.e6. doi: 10.1016/j.cgh.2024.06.004. Epub 2024 Jun 20. PMID 38908733
- [Background] Fang H, Yao T, Li W, Pan N, Xu H, Zhao Q, Su Y, Xiong K, Wang J. Efficacy and safety of fecal microbiota transplantation for chronic insomnia in adults: a real world study. Front Microbiol. 2023 Nov 21;14:1299816. doi: 10.3389/fmicb.2023.1299816. eCollection 2023. PMID 38088972